CLINICAL TRIAL: NCT02182323
Title: Safety, Tolerance, and Pharmacokinetics of Single Oral Doses of 4 mg, 16 mg, 48 mg, 120 mg, 240 mg, 480 mg, 800 mg, and 1200 mg BI 201335 NA (PEG 400/TRIS/Meglumine/Water Solution) in Healthy Male Subjects, in a Randomised Single Blind, Placebo Controlled Rising Dose Study, Followed With an Open-label Intra-subject Two-stage Crossover Pilot Bioavailability Comparison of 480 mg BI 201335 NA in a PEG 400/TRIS/Meglumine/Water Solution Coadministered With Food
Brief Title: Safety, Tolerance, and Pharmacokinetics of Single Oral Doses of BI 201335 NA and Bioavailability in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1220.3
Record Dates: First submitted 2014-07-02; First posted 2014-07-08 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- BI 201335 in single rising doses (Experimental)
  Interventions: Drug: BI 201335 NA
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo solution
- BI 201335 NA fasted or fed (Experimental): two randomized sequences:
  1. BI 201335 NA or placebo fasted
  2. BI 201335 NA or placebo after high-fat breakfast
  Interventions: Drug: BI 201335 NA; Drug: Placebo solution

INTERVENTIONS:
Drug: BI 201335 NA
  Arms: BI 201335 NA fasted or fed; BI 201335 in single rising doses
Drug: Placebo solution
  Arms: BI 201335 NA fasted or fed; Placebo

SUMMARY:
The objective of this study was to investigate the safety, tolerability, and pharmacokinetics of BI 201335 NA following administration of single rising doses from 4 mg to 1200 mg. In addition, the food effect on the bioavailability of BI 201335 NA (480 mg) was investigated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males according to the following criteria: Based upon a complete medical history, including the physical examination, vital signs (Blood Pressure (BP), Pulse Rate (PR)), 12-lead ECG (electrocardiogram), clinical laboratory tests
* Age ≥18 and Age ≤50 years
* BMI ≥18.5 and BMI ≤29.9 kg/m2 (Body Mass Index)
* Signed and dated written informed consent prior to admission to the study in accordance with GCP (Good Clinical Practice) and the local legislation

Exclusion Criteria:

* Any finding of the medical examination (including BP, PR and ECG) deviating from normal and of clinical relevance
* Any evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Prior history of jaundice
* Surgery of the gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
* Intake of drugs with a long half-life (> 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
* Use of drugs which might reasonably influence the results of the trial or that prolong the QT/QTc interval based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
* Participation in another trial with an investigational drug within two months prior to administration or during the trial
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Inability to refrain from smoking alcohol and on trial days
* Alcohol abuse (more than 60 g/day)
* Drug abuse
* Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
* Excessive physical activities (within one week prior to administration or during the trial)
* Any laboratory value outside the reference range that is of clinical relevance
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 ms)
* A history of additional risk factors for TdP (torsade de pointes) (e.g., heart failure, hypokalemia, family history of Long QT Syndrome)

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2006-09; Primary Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Number of patients with abnormal findings in physical examination | up to 12 days
Number of patients with clinically significant changes in vital signs (blood pressure, pulse rate) | up to 12 days
Number of patients with abnormal findings in 12-lead ECG (electrocardiogram) | up to 12 days
Number of patients with abnormal changes in laboratory tests (haematology, clinical chemistry and urinalysis) | up to 12 days
Number of patients with adverse events | up to 12 days
Assessment of tolerability by investigator on a 4-point scale | within 7 days after last trial procedure

SECONDARY OUTCOMES:
Cmax (maximum concentration of the analyte in plasma) | Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 30, 36, 48, 60, 72, 84, 96 hours post-dose
tmax (time from dosing to maximum concentration) | Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 30, 36, 48, 60, 72, 84, 96 hours post-dose
AUC0-infinity (area under the concentration time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 30, 36, 48, 60, 72, 84, 96 hours post-dose
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point) | Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 30, 36, 48, 60, 72, 84, 96 hours post-dose
λz (terminal elimination rate constant in plasma) | Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 30, 36, 48, 60, 72, 84, 96 hours post-dose
t1/2 (terminal half-life of the analyte in plasma) | Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 30, 36, 48, 60, 72, 84, 96 hours post-dose
MRTpo (Mean residence time of the analyte in the body after oral administration) | Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 30, 36, 48, 60, 72, 84, 96 hours post-dose
CL/F (apparent clearance of the analyte in the plasma after oral administration) | Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 30, 36, 48, 60, 72, 84, 96 hours post-dose
Vz/F (apparent volume of distribution during the terminal phase λz following an oral dose) | Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 30, 36, 48, 60, 72, 84, 96 hours post-dose
Aet1-t2 (amount of analyte that is eliminated in urine from the time point t1 to time point t2) | Pre-dose and 0-4, 4-12, 12-24, 24-48 hours post-dose in the single rising dose phase
fet1-t2 (fraction of analyte eliminated in urine from time point t1 to time point t2) | Pre-dose and 0-4, 4-12, 12-24, 24-48 hours post-dose in the single rising dose phase
CLR,t1-t2 (renal clearance of the analyte from the time point t1 until the time point t2) | Pre-dose and 0-4, 4-12, 12-24, 24-48 hours post-dose in the single rising dose phase